CLINICAL TRIAL: NCT04467502
Title: Virtual Reality Exposure Therapy for Gambling Disorder: Randomized Controlled Trial
Brief Title: Virtual Reality Exposure Therapy for Gambling Disorder
Acronym: VIRET-GAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020_02; 2020-A02710-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-06-29; First posted 2020-07-13 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Gambling Disorder
Keywords: Exposure therapy; virtual reality; cognitive behavioral therapy; pathological gambling; CBT
MeSH Terms: conditions — Gambling | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT with VRET (Experimental)
  Interventions: Other: cognitive-behavioral therapy for gambling disorder; Other: virtual reality exposure therapy focus on gambling cues
- CBT with imaginal ET (Active Comparator)
  Interventions: Other: cognitive-behavioral therapy for gambling disorder; Other: imaginal exposure therapy focus on gambling cues

INTERVENTIONS:
Other: cognitive-behavioral therapy for gambling disorder — 6 sessions of cognitive-behavioral therapy for gambling disorder
Other: imaginal exposure therapy focus on gambling cues — 6 sessions of imaginal exposure therapy focus on gambling cues
  Arms: CBT with imaginal ET
Other: virtual reality exposure therapy focus on gambling cues — 6 sessions of virtual reality exposure therapy focus on gambling cues
  Arms: CBT with VRET

SUMMARY:
Gambling disorder (GD) is recognized as an addictive disorder in the DSM-5. Craving is a core phenomenon in addiction that can lead to relapse in problem gambling for pathological gamblers. Exposure Therapy (ET) focuses on craving in addiction treatment. ET in Cognitive-Behavioral Therapy (CBT) is based on classical conditioning that addresses the association between contextual cues and the craving response. ET helps the patient to reduce craving when faced with cues triggering craving. ET includes in vivo exposure and imaginal exposure. The literature recommends being as close as possible to the context of addiction to facilitate the extinction of craving but in vivo ET is complicated to perform. For GD, in outpatient consultation, bringing a patient to a casino presents obstacles (e.g., time, human and financial cost, agreement with casino for therapy).

The study will be to assess the effectiveness of Virtual Reality Exposure Therapy (VRET) in a virtual gambling environment. Various trials show that VRET is no more or less effective than classical ET in CBT but has other advantages for motivation to treatment. This research aims to compare efficacy between CBT with VRET and CBT with imaginal exposure for treatment of GD in a multicenter, randomized, controlled, non-inferiority clinical trial.

DETAILED DESCRIPTION:
Main aim:

Show, within patients seeking care for GD, that VRET integrated with CBT is non-inferior to imaginal ET integrated with CBT on GD symptom reduction at the end of 12 treatment sessions.

Secondary objectives:

1. Show that VRET integrated with CBT is non-inferior to imaginal ET integrated with CBT on GD symptom reduction during the first 12 months post-treatment.
2. Compare the effect of the two therapeutic strategies on GD symptoms (measured by complementary assessments to that used in the main aim), at the end of treatment and during the first 12 months post-treatment.
3. Show the efficacy of VRET integrated with CBT compared to imaginal ET integrated with CBT on gambling behavior, craving, and gambling-related cognitions at the end of treatment and during the first 12 months post-treatment.
4. Show the efficacy of VRET integrated with CBT compared to imaginal ET integrated with CBT on the evolution of anxiety and depressive symptoms at the end of treatment and during the first 12 months post-treatment.
5. Compare the quality of the two therapeutic strategies at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Seek treatment for GD within one of health care facilities participating in the research (first request for treatment and not patients already receiving treatment for gambling disorder in the care center).
* Meet a current diagnosis of gambling disorder according to DSM-5 criteria and with a South Oaks Gambling Screen (SOGS) score ≥ 5
* Meet a casino gambling behavior with a casino gambling frequency ≥ 1 time every two months during the last 12 months
* Have a sufficient understanding of French for therapy
* Beneficiary of the French social security system
* Give an informed consent to participate
* Willing to comply with all study procedures and duration

Exclusion Criteria:

* Visual disturbance making impossible the use of virtual reality equipment (e.g. advanced retinal degeneration, central scotoma, age-related macular degeneration)
* Pregnant woman
* Minor or adult under guardianship, conservatorship, under judicial protection, persons deprived of their liberty
* Balance disorder (e.g. cerebellar disorder, inner ear disorder)
* Photosensitive epilepsy
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in South Oaks Gambling Screen (SOGS) between baseline and end of treatment (12 sessions, 6 months) | at the end of treatment (an average of 6 months)
  The SOGS is a 20-item instrument used to screen for pathological gambling. The SOGS is scored by summing the number of items endorsed out of 20 and a cut score of 5 or more indicates a probable pathological gambling. The score ranges from 0 to 20.

SECONDARY OUTCOMES:
Change in South Oaks Gambling Screen (SOGS) between baseline and follow-up at 3, 6 and 12 months after the end of treatment | at baseline, and through study completion, an average of 18 months
  The SOGS is a 20-item instrument used to screen for pathological gambling. The SOGS is scored by summing the number of items endorsed out of 20 and a cut score of 5 or more indicates a probable pathological gambling. The score ranges from 0 to 20.
Change in gambling disorder symptoms between baseline, end of treatment and follow-up assessed by the following criteria: number of DSM-5 criteria for GD | at baseline, and through study completion, an average of 18 months
  Nine criteria for gambling disorder are described in DSM-5. The endorsement of 4-5 criteria means the presence of a mild gambling disorder, 6-7 criteria a moderate gambling disorder and 8-9 criteria a severe gambling disorder. The score ranges from 0 to 9 criteria.
Change in gambling disorder symptoms between baseline, end of treatment and follow-up assessed by the following criteria: Problem Gambling Severity Index (PGSI) | at baseline, and through study completion, an average of 18 months
  The PGSI consists of nine items to assess level of risk for problem gambling. Cut-off scores are 1-2 for low-risk gamblers, 3-7 for moderate-risk gamblers and 8 or more for problem-gamblers. Non-problem gamblers correspond to 0. The score ranges from 0 to 27.
Change in gambling behavior assessed by gambling frequency during the last month | at baseline, and through study completion, an average of 18 months
Change in gambling behavior assessed by amount of money spent in gambling during the last month | at baseline, and through study completion, an average of 18 months
Change in gambling behavior assessed by time spent gambling during the last month | at baseline, and through study completion, an average of 18 months
Change in frequency subscale of gambling Craving Experience Questionnaire (g-CEQ) | at baseline, and through study completion, an average of 18 months
  The frequency subscale of gambling Craving Experience Questionnaire assesses the frequency of craving for gambling during the last week. This questionnaire consists of nine items. A high score means a high frequency of craving during the last week. The score ranges from 0 to 90.
Change in craving reactivity to gambling cues | at baseline, and through study completion, an average of 18 months
Number of craving episodes using daily craving assessed by participants | up to 6 months during the treatment
Cumulative duration of craving episodes using daily craving assessed by participants | up to 6 months during the treatment
Change in gambling-related cognitions assessed by Gambling-Related Cognitions Scale (GRCS) | at baseline, and through study completion, an average of 18 months
  The French version of the Gambling-Related Cognitions Scale consists of 23 items to assess various cognitions related to gambling. A high score means that gambling-related cognitions are typical cognitions of problem gamblers. The score ranges from 23 to 161.
Change in depressive symptoms assessed by Beck Depression Inventory short-form (BDI-SF) | at baseline, and through study completion, an average of 18 months
  Beck Depression Inventory short-form consists of 13 items to assess depressive symptoms. A high score means a high level of depressive symptoms. The score ranges from 0 to 39.
Change in anxiety symptoms assessed by State-Trait Anxiety Inventory (STAI) | at baseline, and through study completion, an average of 18 months
  State-Trait Anxiety Inventory consists of 20 items to assess state-anxiety and 20 items to assess trait-anxiety. A high score means a high level of anxiety symptoms. The score ranges from 20 to 80 both for state-anxiety and trait-anxiety.
Rate of patients who attended the 12 sessions (6 months) | up to 6 months during the treatment
  Quality of the two therapeutic strategies

CONTACTS AND LOCATIONS:
Overall Officials: Pierre TAQUET, PhD, Principal Investigator — University Hospital, Lille
Locations (10):
- France (10):
  - CHU Amiens-Picardie, Amiens
  - CH Boulogne sur mer CSAPA, Boulogne-sur-Mer
  - CHU de Caen, Caen
  - Hôpital Fontan, CHU lille, Lille
  - Assoriation Cédragir Lomme CSAPA, Lomme
  - CH de l'arrondissement de Montreuil / CSAPA, Montreuil-sur-Mer
  - CHU Rouen, Rouen
  - CH de Saint Amand les Eaux, Saint-Amand-les-Eaux
  - CH Seclin Carvin CSAPA, Seclin
  - Association GREID ValenciennesCSAPA, Valenciennes